CLINICAL TRIAL: NCT04626505
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Reduction in Inflammation in Patients With Advanced Chronic Renal Disease Utilizing Antibody-Mediated Interleukin-6 Inhibition in Japan
Brief Title: Trial to Evaluate Reduction in Inflammation in Patients With Advanced Chronic Renal Disease Utilizing Antibody Mediated IL-6 Inhibition in Japan.
Acronym: RESCUE-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Collaborators: Sponsor: Corvidia Therapeutics Inc, a subsidiary of Novo Nordisk A/S (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6018-4776; U1111-1260-3695 (Other: World Health Organization (WHO)); jRCT2031200216 (Registry Identifier: JAPIC/jRCT)
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Chronic Kidney Disease; Inflammation; Cardiovascular Risk
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — ziltivekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ziltivekimab 15 mg (Experimental): Participants will receive ziltivekimab 15 mg for 12 weeks.
  Interventions: Drug: Ziltivekimab
- Ziltivekimab 30 mg (Experimental): Participants will receive ziltivekimab 30 mg for 12 weeks.
  Interventions: Drug: Ziltivekimab
- Placebo (ziltivekimab) (Placebo Comparator): Participants will receive placebo (ziltivekimab) for 12 weeks.
  Interventions: Drug: Placebo (ziltivekimab)

INTERVENTIONS:
Drug: Ziltivekimab — Administered subcutaneously (s.c., under skin) once every 4 weeks for 12 weeks
  Arms: Ziltivekimab 15 mg; Ziltivekimab 30 mg
Drug: Placebo (ziltivekimab) — Administered s.c. once every 4 weeks for 12 weeks
  Arms: Placebo (ziltivekimab)

SUMMARY:
The purpose of this research study is to compare the safety and effectiveness of 2 different doses of a study drug called ziltivekimab to placebo (an inactive substance) in reducing inflammation and improving some of the bad effects of inflammation on heart disease. Participants will be randomly (by chance) assigned to receive either ziltivekimab or placebo. The chance that participants will be assigned into one of the three study arms of ziltivekimab (either 15 mg or 30 mg) or placebo is the same (approximately 33%). This is a double-blind study, which means neither participants nor the study doctor will know which group the participants are in. In case of an emergency, however, the study doctor can get this information. The study drug will be injected under the skin once every 4 weeks. In this study participants will receive 3 injections of study drug. The total study duration for each participant will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 20 years at the time of signing the Informed Consent Form
* Stage 3 to 5 non-dialysis-dependent chronic kidney disease (NDD-CKD), ie, estimated glomerular filtration rate above 10 and below 60 mL/min/1.73 m^2 using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) creatinine equation
* Serum hs-CRP level equal to or above 2.0 mg/L measured during the screening period. Note: Targeting patients with a history of advanced stage CKD, atherosclerotic cardiovascular disease, anemia, diabetic retinopathy, obesity, or elevated BMI, and diabetes for screening will help increase the chances of identifying patients with hs-CRP equal to or above2.0 mg/L 4. The patient agrees to comply with
* The patient agrees to comply with the contraception and reproduction restrictions of the study as follows:

  1. Women of childbearing potential must be using a method of contraception that is "highly effective" (ie, less than 1% failure rate) for at least 3 months following the last dose of study drug;
  2. Postmenopausal women must have had no menstrual bleeding for at least 1 year before initial dosing and either be over the age of 60 years or have an elevated plasma follicle stimulating hormone level (ie, above 40 mIU/mL) at screening;
  3. Women of childbearing potential must have a documented negative serum pregnancy test result at screening; and
  4. All male patients, from the day of dosing until the final study visit, unless surgically sterile, must be willing to use a condom with a partner (male patients with partners of childbearing potential must be willing to use 2 effective methods of birth control, 1 should be condom with spermicide) to prevent pregnancy and drug exposure of a partner, and refrain from donating sperm or fathering a child; and
* The patient must be willing and able to provide informed consent and abide all study requirements and restrictions.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation in the study:

Laboratory values

* Absolute neutrophil count below 2.0 × 10^9/L during screening;
* Platelet count below 120 × 10^9/L during screening;
* Spot urine protein-creatinine ratio above 4000 mg/g (4.0 g/g) during screening;
* Alanine aminotransferase or aspartate aminotransferase above 2.5 × upper limit of normal during screening;
* Positive testing for tuberculosis during screening. blood testing (eg, QuantiFERON) is preferred, but a purified protein derivative (PPD) skin test read within 48 to 72 hours by a qualified healthcare professional may also be performed. If a patient is PPD positive but QuantiFERON negative, the patient is eligible;
* Evidence of human immunodeficiency virus (HIV)-1 or HIV-2 infection by serology measured during screening;
* Hepatitis B or C by serology (eg, hepatitis B surface antigen or hepatitis C antibody positive) measured during screening;

Medical conditions or diseases

* Expected to require blood transfusion within 12 weeks post-randomization;
* Thromboembolic event within 12 weeks prior to randomization;
* Clinical evidence or suspicion of active infection;
* History of peptic ulcer disease or gastrointestinal ulceration in the 12 months prior to randomization;
* History of active diverticulitis in the 12 months prior to randomization;
* History of inflammatory bowel disease that has been clinically active during the 12 months prior to randomization;
* Uncontrolled hypertension (defined as an average systolic blood pressure above 160 mmHg or an average diastolic blood pressure above 100 mmHg) during screening. Patients may be re-evaluated within 2 weeks, at the discretion of the Principal Investigator, for this criterion if antihypertensive therapy has been started or increased as a result of initial screening blood pressure being above these limits;
* Planned coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) or any other major surgical procedure during the time frame of the study;
* Major cardiac surgical, non-cardiac surgical, or major endoscopic procedure within the past 6 months prior to randomization;
* Prior gastric bypass surgery;
* History of New York Heart Association (NYHA) Class IV congestive heart failure within 12 weeks prior to randomization;
* Diagnosis of malignancy within 1 year prior to randomization with the exception of successfully treated nonmetastatic basal cell or squamous cell carcinomas of the skin and/or local carcinoma in situ of the cervix;
* History of bone marrow or solid organ transplant or anticipated to receive an organ transplant during the time frame of the study;
* Known allergy to the study drug or any of its ingredients;

Prior or current medications

* Received an investigational drug within 30 days prior to screening;
* Received a live vaccine product within 14 days of study drug administration or expect to receive live vaccine during the treatment period;
* Expected to receive any investigational drug or any of the exclusionary drugs during the treatment period or safety follow-Up period;
* Chronic use of systemic immunosuppressive drugs during the screening period or anticipated use of such drugs any time during the study. Note: Use of otic, ophthalmic, inhaled, and topical corticosteroids or local corticosteroid injections are not exclusionary. Oral prednisone up to 5 mg per day (or equivalent) is permitted if the dose has been stable for at least 4 weeks prior to Screening and no dose changes are planned during study participation. Short-term use of oral steroids for treatment of rash or asthma exacerbation is allowed;
* Use of systemic antibiotics, systemic antivirals, or systemic antifungals during the screening period. Note: "Systemic" is defined as oral or intravenous drugs that are absorbed into the circulation;
* Requirement of an indwelling catheter of any type; 28. Use of hypoxia-inducible factor (HIF) stabilizers or erythropoiesis-stimulating agents (ESA) within 6 weeks of randomization or during the treatment period;

General exclusions

* Currently breastfeeding; or
* Any condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or interpretation of the study results, or that would in the opinion of the Investigator increase the risk of participating in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
The difference in the percent change in high-sensitivity C-reactive protein (hs-CRP) levels (average of all hs-CRP values prior to the administration of study drug) between each active group and placebo | From baseline (week 0) to the end of treatment (week 12)
  Percent change

SECONDARY OUTCOMES:
Number of adverse events (AEs) | From randomisation (week 0) to week 20
  Count of events
Number of serious adverse events (SAEs) | From randomisation (week 0) to week 20
  Count of events
Participants with AEs leading to discontinuation | From randomisation (week 0) to week 20
  Count of participant

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Ehime, Japan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Wada Y, Jensen C, Meyer ASP, Zonoozi AAM, Honda H. Efficacy and safety of interleukin-6 inhibition with ziltivekimab in patients at high risk of atherosclerotic events in Japan (RESCUE-2): A randomized, double-blind, placebo-controlled, phase 2 trial. J Cardiol. 2023 Oct;82(4):279-285. doi: 10.1016/j.jjcc.2023.05.006. Epub 2023 May 19. PMID 37211246